CLINICAL TRIAL: NCT02471703
Title: Clinical Outcome Following Total Hip Arthroplasty With the SMF Stem A Prospective, Consecutive Series, Multi-center Clinical Study
Brief Title: Clinical Outcome Following Total Hip Arthroplasty With the SMF Stem
Acronym: SMF-S&E
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely terminated by S+N due to business reasons. After an extensive review of all ongoing studies with the focus on which studies are still required for regulatory obligations S+N took the decision to close the SMF S&E study.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011SMFH132_R11007-1
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Joint Diseases
Keywords: Total Hip Arthroplasty; Total Hip Replacement; Inflammatory Joint Disease; Non-Inflammatory Joint Disease
MeSH Terms: conditions — Joint Diseases | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SMF mini-stem hip replacement recipient: Received the device via total hip arthroplasty
  Interventions: Device: Total hip arthroplasty

INTERVENTIONS:
Device: Total hip arthroplasty — Total hip arthroplasty
  Other Names: Total hip replacement

SUMMARY:
This is a prospective, consecutive series, multicenter clinical study of clinical outcomes following total hip arthroplasty with the SMF stem.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the safety and efficacy of the study device. This study will document any device-related, surgical or post-operative complication and adverse radiographic observations. Improvement in pain, function, and health economic data will be compared with improvements documented with other joint systems. Outcome measures will be quantified through statistical analysis of study device , HOOS questionnaire, radiographic assessments, Harris Hip Score, and adverse event reports.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with non-inflammatory degenerative joint disease including osteoarthritis, traumatic arthritis, avascular necrosis, rheumatoid arthritis of or any of it's composite diagnosis.
* Patient is of legal age to consent, is skeletally mature and at least 18 years old.
* Patient is willing to consent to participate in the study by signing and dating an IRB-approved consent form.
* Patient is in stable health and is free of or treated and stabilized for cardiac, pulmonary, hematological or other conditions that would pose excessive operative risk.

Exclusion Criteria:

* Patient has poor bone stock and would make the procedure unjustifiable: A) patients which are under medical care for osteoporosis (taking hormones, Calcitonin or biphosphates) or for other metabolic pathologies, which could influence the quality of the bone (for example hyperparathyroidism, hyperthyreoidismus and osteomalacie) will be excluded from the study. B) patients suffering from Morbus Paget (osteodystrophia deformans) will be excluded from the study.
* Patient has conditions that tend to place increased loads on implants such as weight, chargot joint, muscular deficiencies and activity level, which are incompatible with a satisfactory long-term result: A) patients with a BMI > 40 will be excluded from the study B) patients participating in high-impact sports like baseball, basketball, football, handball, hockey, karate, racquet-ball, running, soccer, water skiing or similar impact sports will be excluded from the study.
* Patient is over the age of 75.
* Skeletal immaturity: patients must be at least 18 years at the time of the operation.
* Patient has an active, local infection that would lead to increased bone resorption.
* Mental or neurological conditions that tend to pre-empt the patient's ability or willingness to restrict activities.
* Known sensitivity to materials of the implant.
* Patient is pregnant or plans to be come pregnant during the course of the study.
* Patient is a prisoner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring total hip replacement.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2008-02-27 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Revision of the study device | Discharge through 10 years
  Instances of required revision of the study device
Device related Adverse Events | Implant through 10 years
  surgical, device-related, death and serious adverse events will be analyzed
Harris Hip Score | Baseline through 10 years
  Questionnaire to calculate pain, walking abilities, activities, degrees of hip motion
HOOS Questionnaire | Baseline through 10 years
  Questionnaire to calculate hip symptoms, stiffness, pain, function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Parveen, Study Chair — Smith & Nephew, Inc.
Locations (6):
- ZNA Middleheim, Berchem, Belgium
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Hmr, Montreal, Quebec
  - CHUQ-L'Hôtel-Dieu de Québec, Québec, Quebec
- Germany (2):
  - St. Vincenz Hospital, Brakel
  - Brüderkrankenhaus St. Josef, Paderborn